CLINICAL TRIAL: NCT07154420
Title: Periodontal Status and Quality of Life in Patients With Psoriasis: A Cross-Sectional Study
Brief Title: Periodontal Health and Quality of Life in Psoriasis Patients
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Gülbahar Ustaoğlu, associate professor, Saglik Bilimleri Universitesi
Other Study IDs: GUSTAOGLU
Record Dates: First submitted 2025-08-19; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Psoriasis; Periodontal Diseases
Keywords: psoriasis,periodontitis
MeSH Terms: conditions — Psoriasis; Periodontal Diseases; Periodontitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- psoriasis patient group
  Interventions: Diagnostic Test: Diagnostic Test: Periodontal Examination
- healthy control group
  Interventions: Diagnostic Test: Diagnostic Test: Periodontal Examination

INTERVENTIONS:
Diagnostic Test: Diagnostic Test: Periodontal Examination — Diagnostic Test: Periodontal Examination
Diagnostic Test: Diagnostic Test: Periodontal Examination — Periodontal Examination

SUMMARY:
This study aims to evaluate the relationship between psoriasis, a chronic inflammatory skin disease, and oral health. We will assess the periodontal (gum) condition of patients with psoriasis and examine how it affects their quality of life. A group of psoriasis patients and a control group without psoriasis will undergo oral examinations and complete a short questionnaire. The goal is to better understand whether psoriasis has an impact on gum health and daily well-being.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 65 years
* Clinically diagnosed with active psoriasis
* The presence of at least 12 teeth (excluding third molars)
* Absence of contraindications for periodontal clinical examination

Exclusion Criteria:

* Other dermatological conditions
* Pregnancy or lactation
* Antibiotic use within the last 3 months
* Chemotherapy or radiotherapy within the last year
* Periodontal treatment within the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants aged 18 to 65 years, clinically diagnosed with active psoriasis, and applying to the Dermatology and Venereal Diseases Department outpatient clinic of the Gulhane Faculty of Medicine were recruited into the test group (n=113). The control group consisted of healthy individuals without any dermatological or systemic diseases (n=113).
Sampling Method: Non-Probability Sample
Enrollment: 226 (Actual)
Dates: Start 2025-04-20 (Actual); Primary Completion 2025-07-20 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of oral health-related quality of life in psoriasis patients | Baseline
  The Turkish version of the OHIP-14 questionnaire was administered through face-to-face interviews by a single investigator (G.U.), who was blinded to the periodontal status of the participants. The OHIP-14 consists of seven subscales, each including two items: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and handicap. Participants rated the frequency of negative experiences on a five-point Likert scale (0 = never, 1 = rarely, 2 = occasionally, 3 = quite often, 4 = very often). The total score ranges from 0 to 56, with higher scores reflecting a greater negative impact on oral health-related quality of life

SECONDARY OUTCOMES:
Evaluation of dermatology-specific quality of life in psoriasis patients | Baseline
  Psoriasis Quality of Life Questionnaire (PQLQ) measures functional limitation, physical discomfort, psychological distress, social maladjustment, and disability. Each item was scored on a Likert-type scale, with higher scores reflecting a greater impact on daily life.

CONTACTS AND LOCATIONS:
Locations (1):
- Sağlık Bilimleri Üniversitesi, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No